CLINICAL TRIAL: NCT03791788
Title: Multicenter Registry for Diagnostic Accuracy of Angiography-Derived Quantitative Flow Ratio to Evaluate the Hemodynamic Significance of Coronary Artery Stenosis
Brief Title: Multicenter Registry for Angiography-Derived Quantitative Flow Ratio
Acronym: QFRRegistry
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Collaborators: Seoul National University Hospital (Other); Inje University (Other); Dongsan Medical Center (Other); Chosun University Hospital (Other)
Responsible Party: Principal Investigator, Joo Myung Lee, Assistant Professor, Samsung Medical Center
Other Study IDs: QFR2018-11-112-002
Record Dates: First submitted 2018-12-28; First posted 2019-01-03 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Ischemic Heart Disease
Keywords: Stable angina; Acute Myocardial Infarction; Fractional Flow Reserve; Quantitative Flow Ratio
MeSH Terms: conditions — Myocardial Ischemia; Angina, Stable

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- QFR Group: Patients with suspected ischemic heart disease including stable angina, or acute coronary syndrome including unstable angina, NSTEMI (non ST-segment elevation myocardial infarction), or STEMI (ST-segment elevation myocardial infarction) with non-culprit stenosis who underwent FFR measurement and were able to analyze QFR.
  Interventions: Diagnostic Test: QFR assessment

INTERVENTIONS:
Diagnostic Test: QFR assessment — QFR measurement in order to evaluate functional significance of epicardial stenosis and to compare the response of QFR for worsening stenosis severity, FFR value as reference standard

SUMMARY:
1. to investigate the feasibility and diagnostic performance of contrast quantitative flow ratio (QFR) for identifying the functional significance of intermediate degree stenotic lesions in all-comer patients with coronary artery disease (CAD) including presentation of acute myocardial infarction (AMI) with non-culprit lesion.
2. to compare the changes of contrast QFR and fractional flow reserve (FFR) according to severity of percent diameter stenosis (%DS)
3. to evaluate prognostic implication of contrast QFR in comparison with FFR

DETAILED DESCRIPTION:
Despite potential clinical benefits and abundant evidences of FFR-guided percutaneous coronary intervention (PCI), adoption rate of FFR is still low in real world practice, most likely due to use of additional resource and to concern about side effects of hyperemic agent. Therefore, several tools to derive FFR non-invasively has been developed based on computational fluid dynamics to overcome the limitations. One of the novel methods, the contrast quantitative flow ratio (QFR) is a computation of FFR based on 3-dimensional quantitative coronary angiography (QCA) combined with Thrombolysis in Myocardial Infarction (TIMI) frame counts adjustment without hyperemic agent infusion.

Although diagnostic performance of contrast QFR for evaluation of functional significance, using FFR as reference standard, is well validated in patients with stable ischemic heart disease (SIHD), there have been lack of evidence regarding the reliability of QFR for non-culprit stenosis in patients with AMI.

Therefore, the investigators sought to investigate the feasibility and diagnostic performance of contrast QFR for identifying the functional significance of coronary stenosis in all-comer patients with CAD. In addition, prognostic implication of contrast QFR will be also compared with that of FFR.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be ≥18 years
* Patients suspected with ischemic heart disease
* Patients with intermediate degree of coronary artery stenosis (40-70% stenosis by visual estimation) in major epicardial coronary artery with FFR measurement
* Patients who were able to analyze QFR
* Subject is able to verbally confirm understandings of risks, benefits and treatment alternatives of receiving invasive physiologic evaluation and he/she or his/her legally authorized representative provides

Exclusion Criteria:

* Left main (LM) or right coronary artery (RCA) ostial lesion
* Severe overlap of stenotic segments
* Severe tortuosity of target vessel
* Poor angiographic image quality precluding contour detection
* No optimal images with angles ≥ 25o

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 320 patients with suspected ischemic heart disease including stable angina, or acute coronary syndrome including unstable angina, non ST-segment elevation MI, or ST-segment elevation MI with non-culprit stenosis who underwent FFR measurement and were able to analyze QFR
Sampling Method: Non-Probability Sample
Enrollment: 524 (Actual)
Dates: Start 2016-04-30 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of QFR | through study completion, an average of 6 months
  Diagnostic accuracy of contrast QFR to predict FFR lower than 0.8
Vessel-related composite outcome | through study completion, an average of 2 year
  a composite of cardiac death, vessel-related myocardial infarction, and vessel-related ischemia driven revascularization

SECONDARY OUTCOMES:
Sensitivity of QFR | through study completion, an average of 6 months
  Sensitivity of contrast QFR to predict FFR lower than 0.8
Specificity of QFR | through study completion, an average of 6 months
  Specificity of contrast QFR to predict FFR lower than 0.8
Correlation between QFR and FFR | through study completion, an average of 6 months
  Correlation between QFR and FFR

OTHER OUTCOMES:
Pre-specified substudy of exercise duration after PCI | through study completion, an average of 3 months
  residual functional SYNTAX score calculated using post-PCI QFR will be used to define functional complete revascularization.
  Pre- and Post-PCI exercise treadmill test within 3 months window from PCI

CONTACTS AND LOCATIONS:
Overall Officials: Joo Myung Lee, MD, MPH, PhD, Principal Investigator — Samsung Medical Center
Locations (5):
- South Korea (5):
  - Keimyung University Dongsan Medical Center, Daegu
  - Inje University Ilsan Paik Hospital, Goyang-si
  - Chosun University Hospital, Gwangju
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul